CLINICAL TRIAL: NCT01912014
Title: Psychosocial Wellbeing Following Stroke: Developing and Testing a Psychosocial Nursing Intervention for Primary Care
Brief Title: Psychosocial Wellbeing Following Stroke
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Marit Kirkevold, Professor, University of Oslo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2.2007.37 (REK); 16369 (Social science data)
Record Dates: First submitted 2013-07-24; First posted 2013-07-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Psychosocial; Narrative; Coping; Quality of Life
Keywords: stroke; psychosocial; intervention; quality of life
MeSH Terms: conditions — Narration; Stroke | interventions — Psychiatric Rehabilitation; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Psychosocial support and counselling (Experimental): There is only one arm as this is a pilot and feasibility study.
  Interventions: Behavioral: Psychosocial support and counselling

INTERVENTIONS:
Behavioral: Psychosocial support and counselling

SUMMARY:
The purpose of this feasibility study is to develop and initially test a dialogue-based psychosocial intervention aimed at promoting coping and psychosocial wellbeing following an acute stroke. The intervention is carried out by primary care registered nurses or other appropriate health professionals. The intervention included persons with and without aphasia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or above
* acute stroke
* 4-8 weeks poststroke

Exclusion Criteria

* Other serious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-01; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Stroke and Aphasia Quality of Life (SAQOL-39) | baseline and 2 weeks after end of intervention

SECONDARY OUTCOMES:
Change from baseline in Stroke and Aphasia Quality of Life (SAQOL-39) | baseline and 12 months after end of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Background] Kirkevold M, Bronken BA, Martinsen R, Kvigne K. Promoting psychosocial well-being following a stroke: developing a theoretically and empirically sound complex intervention. Int J Nurs Stud. 2012 Apr;49(4):386-97. doi: 10.1016/j.ijnurstu.2011.10.006. Epub 2011 Nov 1. PMID 22051438
- [Result] Bronken BA, Kirkevold M. Between the lines: generating good qualitative data in studies involving persons with aphasia. ANS Adv Nurs Sci. 2013 Apr-Jun;36(2):E14-28. doi: 10.1097/ANS.0b013e318290200a. PMID 23644268
- [Result] Bronken BA, Kirkevold M, Martinsen R, Wyller TB, Kvigne K. Psychosocial well-being in persons with aphasia participating in a nursing intervention after stroke. Nurs Res Pract. 2012;2012:568242. doi: 10.1155/2012/568242. Epub 2012 Jul 22. PMID 22888417
- [Derived] Kirkevold M, Martinsen R, Bronken BA, Kvigne K. Promoting psychosocial wellbeing following stroke using narratives and guided self-determination: a feasibility study. BMC Psychol. 2014 Feb 3;2(1):4. doi: 10.1186/2050-7283-2-4. eCollection 2014. PMID 25566379